CLINICAL TRIAL: NCT00334659
Title: A Double-blind, Placebo-controlled, Positive Controlled, Randomized, Crossover Study to Investigate the Cardiovascular Safety of Apricitabine in Healthy Subjects
Brief Title: A Study to Investigate the Cardiovascular Safety of Apricitabine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avexa (Industry)
Responsible Party: Susan Cox, Avexa
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: AVX-101
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV-1 Infection
MeSH Terms: conditions — HIV Infections | interventions — apricitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: apricitabine

SUMMARY:
The purpose of this study is to confirm that apricitabine does not induce any clinically significant effect upon electrocardiogram (ECG) parameters at doses consistent with the maximum exposure expected to occur in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18 - 65 years of age, inclusive.
* Body mass index (BMI) between 18-30 kg/m2, inclusive, and a total body weight > 50 kg.
* No clinically significant medical history.
* No clinically significant findings on complete physical examination, including blood pressure, pulse rate and 12-lead ECG.
* Normal clinical safety laboratory results at screening.
* Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.
* Willing and able to stay in the clinic for the in-patient activities required by the protocol.

Exclusion Criteria:

* Evidence of clinically relevant pathology that could interfere with the study results or put the subject's safety at risk.
* Current or recurrent disease that may affect the action, absorption or disposition of the study treatment, or clinical or laboratory assessments.
* Current or relevant previous history of serious, severe or unstable (acute or progressive) physical or psychiatric illness, any medical disorder requiring treatment or that may make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study treatment or procedures.
* History of febrile illness within the 5 days prior to the first dose.
* Positive Hepatitis B surface antigen, Hepatitis C antibody or HIV test result at screening visit.
* Use of any prescription medication within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication or during the study. As an exception, acetaminophen may be used at doses of ≤ 1 g/day.
* Use of any over-the-counter (OTC) medication within 7 days or 5 half-lives (whichever is longer) prior to or during the study. Herbal supplements (including herbal weight-loss or "metabolism booster" therapies) must be discontinued 28 days prior to the first dose of trial medication.
* Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds or any of their stated ingredients.
* Subjects with a history of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces [150 ml] of wine, 12 ounces [360 ml] of beer or 1.5 ounces [45 ml] of hard liquor) or illicit substance abuse within 6 months of screening.
* Positive screen for alcohol or drugs of abuse during screening visit or at study check-in.
* History or evidence of routine use of tobacco or nicotine-containing products in excess of 5 cigarettes per day (or equivalent).
* Participated in a clinical study involving an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
* Blood donation of one pint or more within 56 days of the start of the study.
* Plasmapheresis or plasma donation within 30 days of the start of the study.
* Single 12-lead ECG demonstrating QTc > 450 msec at screen. A single repeat ECG may be done at the investigator's discretion.
* Any condition that in the opinion of the investigator would complicate or compromise the study, or the well-being of the subject.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
QTc at individual Day 7 post-dose Tmax as determined by concurrent pharmacokinetic (PK) analysis for apricitabine | day 7
The maximum Day 7 QTc increase from baseline observed between 1 to 4 hours post-dose, using time-matched ECG assessments | day 7
The average Day 7 QTc observed between 1 to 4 hours post-dose | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Cox, PhD, Study Director — Avexa
Locations (1):
- Jasper Clinic Inc., Kalamazoo, Michigan, United States